CLINICAL TRIAL: NCT03497923
Title: Interaction Between Intravenous Magnesium Sulphate and Neostigmine or Sugammadex for the Reversal of a Rocuronium-induced Neuromuscular Block - A Randomized, Double Blinded, Electrophysiological Study
Brief Title: Interaction Between Magnesium and Neostigmine or Sugammadex for the Reversal of a Rocuronium-induced Neuromuscular Block
Acronym: MagNeoSug
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christoph Czarnetzki (Other)
Collaborators: Hôpital du Valais (Other)
Responsible Party: Sponsor-Investigator, Christoph Czarnetzki, Doctor, MBA, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCER 2016-00018
Record Dates: First submitted 2017-12-26; First posted 2018-04-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Neuromuscular Blockade
Keywords: rocuronium, magnesium sulphate, neostigmine, sugammadex
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: 2 arms, randomized, double blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine (Active Comparator): Patients are anesthesized with Propofol and receive 0.6mg-1 of rocuronium for tracheal intubation. Neuromuscular monitoring will be done on the ulnar nerve by train-of-four (TOF) using a TOF-Watch-SX® acceleromyograph (Organon [Ireland] Ltd). After spontaneous recovery of 2 twitches at the train-of-four monitor (TOF), patients receive neostigmine 50 μg kg-1.
  Interventions: Drug: Magnesium Sulfate
- Sugammadex (Experimental): Patients are anesthesized with Propofol and receive 0.6mg-1 of rocuronium for tracheal intubation. Neuromuscular monitoring will be done on the ulnar nerve by train-of-four (TOF) using a TOF-Watch-SX® acceleromyograph (Organon [Ireland] Ltd). After spontaneous recovery of 2 twitches at the train-of-four monitor (TOF), patients receive sugammadex (Bridion®) 2 mg kg-1.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — After reversal the obention of a TOF ratio of 0.9 is avaited. 10 minutes later patients will receive a perfusion of magnesium 60 mg kg-1 over 5 minutes.

SUMMARY:
Magnesium sulphate is regularly used in perioperative medicine. During and after general anesthesia, it enhances the effect of muscle relaxants because it reduces the liberation of acetylcholine at the neuromuscular junction. When administered immediately after spontaneous recovery of a neuromuscular block (NMB), magnesium may cause a recurrence of NMB and compromise patient safety.

Rocuronium is a neuromuscular blocking agent which is frequently used to facilitate intubating and surgical conditions. At the end of the procedure, there are two ways to accelerate the reversal of a neuromuscular block induced by rocuronium: 1. Administration of neostigmine, an anticholinesterase agent and competitive antagonist; 2. Administration of sugammadex, a γ-cyclodextrin compound and specific encapsulator of rocuronium.

The study is done in patients receiving rocuronium and either neostigmine or sugammadex for reversal of NMB. It is hypothesized that when sugammadex is used as an antagonist of a rocuronium-induced NMB, it prevents the reappearance of NMB when magnesium is injected, because sugammadex should inactivate all remaining rocuronium molecules and restore neuromuscular reserve of the neuromuscular junctions. Further more it is hypothesized that reversal with neostigmine will not prevent a magnesium-induced recurrence of NMB to the same extent. The primary objective of the study is to show that after reversal with sugammadex there is no or only very little re-occurrence of neuromuscular block after a magnesium perfusion. Furthermore we want to show that after reversal with neostigmine there is a re-occurrence of neuromuscular block.

DETAILED DESCRIPTION:
Magnesium sulphate (MgSO4) is regularly used in perioperative medicine. For instance, pre-eclampsia and eclampsia have been successfully treated with intravenous magnesium. Also, MgSO4 has been used for the control of life threatening cardiac arrhythmias, bronchial asthma or as an anticonvulsant. Finally, magnesium has been found to alleviate postoperative pain and to exert morphine sparing effect.

Magnesium plays a role in nearly every physiological system. In the nervous system, magnesium has a depressant effect related to the inhibition of transmitter release from presynaptic sites by competing with calcium and due to the antagonism at NMDA receptors. The presynaptic inhibition of acetylcholine release at the neuromuscular junction by magnesium has been well described. In addition, an excess of magnesium ions diminishes the depolarizing action of acetylcholine at the end-plate, and depresses the excitability of the muscle fiber membrane. Magnesium per se causes significant neuromuscular blockade (NMB) in high concentrations (≥ 5 mmol L-1). In the presence of curare-like agents, however, very low concentrations of magnesium (≥1 mmol L-1) inhibit neuromuscular transmission since in this case much more acetylcholine is needed to produce a magnitude of depolarization of the end-plate compared with normal conditions. Consequently, magnesium enhances the effect of muscle relaxants during and after general anesthesia. The prolongation of the duration of NMB by magnesium may increase the incidence of a residual postoperative neuromuscular block, and consequently may compromise patient safety. In addition, magnesium, when administered immediately after spontaneous recovery of a NMB, may cause recurrence of the NMB ("recurarisation"). Under clinical conditions this may happen whenever magnesium is used in the immediate postoperative period, for instance, for postoperative pain alleviation or for treatment of postoperative cardiac arrhythmia.

It is not known, however, whether pharmacological reversal of a NMB prior to magnesium treatment prevents the recurrence of NMB. Recovery after neostigmine (an anticholinestherase agent) administration was approximately 30% less in patients pretreated with MgSO4 compared with those without MgSO4 pretreatment. Sugammadex, a γ-cyclodextrin compound, is a new reversal agent. It is a specific encapsulator of steroidal muscle relaxants such as rocuronium. We have demonstrated that magnesium pretreatment did not prolong the reversal of deep or moderate rocuronium-induced neuromuscular blockade when standard doses of sugammadex were used for reversal.

Sugammadex causes a rapid and complete reversal of the neuromuscular blockade by reducing the action of rocuronium on the prejunctional and postjunctional nicotinic acetylcholine receptors (nAChRs). Unlike neostigmine, sugammadex is efficacious in reversing moderate (2 twitches to train-of-four [TOF] stimulation, TOF-count two [TOFC-2]) and deep (post-tetanic count [PTC] of 1 or 2) rocuronium-induced NMB in doses of 2.0 mg kg-1 and 4.0 mg kg-1, respectively.

The suggested cause of return of NMB ("recurarisation") subsequent to magnesium administration is the absence of a functional reserve of the neuromuscular junction (safety margin, 70% of receptor capacity) despite a complete recovery of the TOF ratio and twitch amplitude (T1) (main variables of neuromuscular monitoring). It is important to know that the actually available neuromuscular monitoring methods are insensitive to measure the safety margin of the neuromuscular transmission, thus they cannot provide information about the likelihood of block recurrence. Theoretically, recurrence of a NMB due to clinical doses of magnesium happens only in cases where the safety margin is reduced or abolished by a NMB agent. Therefore, to prevent recurrent muscle weakness ideally all relaxant molecules should be eliminated from the neuromuscular synapse before magnesium is administered.

Pharmacological reversal of NMB reduces neuromuscular receptor occupancy and thereby increases the safety margin. Neostigmine augments the amount of acetylcholine at the neuromuscular junction, which competitively antagonizes the NMB and liberates at least partially the synaptic receptor reserves. However, neostigmine is not reliable to completely re-establish neuromuscular function. When sugammadex is administered, the free rocuronium plasma concentration rapidly declines near to zero (like a washout) and consequently the safety margin isincreased. In this context, one can speculate that sugammadex is an ideal antagonist when magnesium treatment is associated with the use of rocuronium.

However, it is still unknown whether the administration of magnesium sulphate immediately after pharmacological reversal of the TOF ratio to a normalized 0.9 value (i.e. adequate reversal) re-induces a clinically relevant NMB. If magnesium is used in the immediate postoperative period, we need to know whether, and how, postoperative muscle paralysis as a consequence of the magnesium treatment can be prevented.

The hypothesis of this study is that when sugammadex is used as an antagonist of a rocuronium- induced NMB, the neuromuscular junction will be liberated from almost all rocuronium molecules and no recurrent NMB will occur. Furthermore it is hypothesized that reversal with neostigmine will not prevent to the same extent magnesium-induced recurrence of NMB. In addition, the magnitude and time course of the magnesium induced neuromuscular block will be measured.

ELIGIBILITY:
Inclusion criteria

Participants fulfilling all of the following inclusion criteria are eligible for the study:

1. Patients, age ≥18 to and ≤ 65 years
2. American Society of Anesthesiology [ASA] status I or II
3. Patient is able to read and understand the information sheet and to sign and date the consent form
4. Patient scheduled of elective surgery lasting ≥100 minutes
5. For women of childbearing age: negative pregnancy test (urinary or blood test)
6. For women of childbearing age: women on the pill should be advised to follow the missed dose advice in the product information; women using non-oral hormonal contraceptives, such as depot formulation, should be advised to use additional contraception for the next seven days

Non-inclusion criteria

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

1. A history of allergy or hypersensitivity to rocuronium, glycopyrronium bromide, neostigmine methylsulfate, sugammadex, or magnesium sulphate
2. Neuromuscular disease receiving medications known to influence neuromuscular function (for instance, aminoglycosides or phenytoine)
3. Preoperative medications known to influence neuromuscular function (for instance aminoglycosides, phenytoin, lidocaine)
4. Patients under toremifene, flucloxacillin and fusidic acid treatment (interaction with sugammadex cannot not be excluded)
5. Documented electrolyte abnormalities (for instance, hypermagnesemia)
6. Documented atrioventricular heart block
7. Patients with magnesium treatment within 3 days before study inclusion
8. Patients with a body mass index <19 or >30 kg/m2
9. Patient having participated in any clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial.
10. Patients undergoing interventions that need a continuous deep NMB (for surgical reasons).
11. Pregnant or breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a decrease in TOF ratio after magnesium administration | Patients will be followed over 24 hours
  Two consecutive measures with a value inferior to TOF 0.9

SECONDARY OUTCOMES:
Lowest TOF ratio measured after starting the magnesium perfusion | 120 minutes
  TOF monitoring every 15 seconds
Time required for the TOF ratio to reach a TOF 0.9 | 120 minutes
  Time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Czarnetzki, MD, MBA, Study Chair — University Hospital Geneve
Locations (2):
- Switzerland (2):
  - University Hospital of Geneva, Anesthesia Department, Geneva, Canton of Geneva
  - Hôpital du Valais, Sion